CLINICAL TRIAL: NCT01151202
Title: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of "AG NPP709 Syrup" in Acute Upper Respiratory Tract Infection and Chronic Inflammatory Bronchitis Patients: Double Blinded, Randomized, Active Drug Comparative, Parallel Designed, Multi-centered, Phase III Study
Brief Title: Therapeutic Confirmatory Clinical Trial to Evaluate the Safety and Efficacy of "AG NPP709 Syrup"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Collaborators: Kyunghee University Medical Center (Other); Inha University Hospital (Other); Ewha Womans University (Other); Hanyang University (Other); Konkuk University Medical Center (Other)
Responsible Party: Jung Hoon, Han, Ahn-Gook Pharmaceutical Co., Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG NPP_P3
Record Dates: First submitted 2010-06-23; First posted 2010-06-28 (Estimated); Last update posted 2010-10-05 (Estimated); Status verified 2010-10

CONDITIONS: Acute Upper Respiratory Tract Infections; Bronchitis
Keywords: acute upper respiratory tract infection, chronic inflamatory bronchitis
MeSH Terms: conditions — Bronchitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AG NPP709 syrup (Experimental): AG NPP709 contains Ivy leaf extract and coptis rhizoma extract
  Interventions: Drug: AG NPP709syrup
- Ivy leaf extract syrup (Active Comparator)
  Interventions: Drug: AG NPP709syrup

INTERVENTIONS:
Drug: AG NPP709syrup

SUMMARY:
The purpose of this study is to assess therapeutic confirmation of AG NPP709 syrup to evaluate the safety and efficacy in patients with acute upper respiratory tract infection and chronic inflammatory bronchitis.

ELIGIBILITY:
Inclusion Criteria:

1. Parent s or patient who decided to participate in this clinical trial at his (her) own will and agreed in written letter of consent
2. Patient ages between 24months and 75years
3. Patient with a clinical diagnosis of acute upper respiratory tract infection or chronic inflammatory bronchitis should has any combination of at least two of following symptoms including sputum: cough, sputum, dyspnea and chest pain when breathing
4. Females of child-bearing age should have nagative pregnancy test or have sufficient contraceptive protection

Exclusion Criteria:

1. Patient whose the following severe respiratory disease: pneumonia, uncontrolled asthma, pancreatic fibrosis viral influenza, tuberculosis
2. Patient whose the following disease: malignant tumors, severe central nervous system disorders, medication needed severe metabolic disorders
3. Patient whose fructose intolerance
4. Patient who has hypersensitivity anamnesis of Prospan syrup
5. Patient whose heart function is abnormal: cardiac insufficiency, including the case of showing abnormal EKG test value that is clinically significant
6. Patient whose liver or kidney function is serious abnormal: including the cases of ALT, AST, bilirubin and blood creatinine value exceeding three times of their upper limit, severe liver disorders, chronic kidney disease
7. Patient who has uncontrolled diabetes or uncontrolled hypertensions
8. Patient who has experience to have participated in other clinical trial within two months before starting the trial
9. Pregnant women, lactating women

Ages: 24 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
improvement by global assessment | 5 days
  At closing visit, researcher assess clinical efficacy using the following five criteria (4: cure, 3: significant improvement, 2: improvement, 1: some improvement, 0: non-improvement or worsening of symptoms). Upper the Grade 3 outcomes are defined as "clinical success".

SECONDARY OUTCOMES:
determine safety by unwanted reaction, clinical laboratory test and physical examination | 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Young-ho Na, PhD, MD, Study Director — Kyung Hee University Medical Center, Department of Pediatrics,
Locations (6):
- South Korea (6):
  - Inha University Hospital, Department of Pediatrics, Incheon
  - Ewha Womens University Medical Center Mokdong Hospital, Department of Allergology, Seoul
  - Hanyang University Medical Center, Department of Respiratory Medicine, Seoul
  - Konkuk University Medical Center, Department of Respiratory Medicine, Seoul
  - Kyung Hee University International Medical Service, Department of Pediatrics, Seoul
  - Kyung Hee University Medical Center, Department of Pediatrics,, Seoul